CLINICAL TRIAL: NCT05077956
Title: Sema 4A as a Marker for Inflammatory Disease in Multiple Sclerosis
Acronym: Sema4A MS
Status: Withdrawn | Type: Observational
Why Stopped: No participants were enrolled before closing the study
Sponsor: Providence Health & Services (Other)
Collaborators: Milton S. Hershey Medical Center (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021000250
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Relapsing Multiple Sclerosis; Multiple Sclerosis
Keywords: multiple sclerosis; relapsing multiple sclerosis; semaphorin 4A; sema4a; disease modifying therapy; biomarker
MeSH Terms: conditions — Multiple Sclerosis; Cone-Rod Dystrophy 10

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sema4A is measured in serum and CSF by a Sema-4A-specific ELISA (Biomatik). Frozen serum and CSF samples will be sent to laboratory at Penn State for these measurements. Whole blood and CSF will be obtained from each subject at the screening/baseline visit, with follow-up whole blood at 6 and 12 months in patient Groups 1-3. We will also measure myelin basic protein levels in the CSF and measure lymphocyte subsets in whole blood for Groups 1-3. These two tests will be performed by the Providence clinical lab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Recently Diagnosed Multiple Sclerosis: Recently diagnosed MS, who have had a clinical attack within the last 6 months, have not received steroids in the last 30 days, and have not started on a disease modifying therapy (DMT).
  Interventions: Diagnostic Test: Cerebrospinal and Blood Serum Semaphorin 4A Levels
- Clinically Stable Relapsing Multiple Sclerosis: Clinically stable relapsing MS, who are receiving a FDA-approved MS DMT and have had no evidence of a clinical relapse for at least the past 12 weeks or gadolinium enhancing lesions on MRI in the prior 4 weeks.
  Interventions: Diagnostic Test: Cerebrospinal and Blood Serum Semaphorin 4A Levels
- Relapsing Multiple Sclerosis on Disease Modifying Therapy: Relapsing MS on a FDA-approved DMT with evidence of recent breakthrough disease, with a documented clinical relapse and/or gadolinium-enhancing lesion(s) on brain or spinal cord MRI taken within the 4 weeks.
  Interventions: Diagnostic Test: Cerebrospinal and Blood Serum Semaphorin 4A Levels
- Healthy Volunteers: Patients without evidence of inflammatory systemic or CNS disease, who require CSF removal for some other cause, such as for idiopathic intracranial hypertension or communicating hydrocephalus.
  Interventions: Diagnostic Test: Cerebrospinal and Blood Serum Semaphorin 4A Levels

INTERVENTIONS:
Diagnostic Test: Cerebrospinal and Blood Serum Semaphorin 4A Levels — Cerebrospinal fluid and serum will be collected at baseline to measure the level of semaphorin 4A.

SUMMARY:
Measure serum and cerebrospinal fluid Sema4A levels in female subjects with newly diagnosed and untreated relapsing multiple sclerosis, clinically stable relapsing multiple sclerosis receiving disease modifying therapy, relapsing multiple sclerosis receiving disease modifying therapy with breakthrough disease, or non-multiple sclerosis controls (patients without inflammatory central nervous system disease).

DETAILED DESCRIPTION:
This pilot study proposal will further investigate whether Semaphorin 4A (Sema4A) elevation in cerebrospinal fluid (CSF) and serum is a potential disease activity biomarker in patients with multiple sclerosis (MS).

A total of 40 female subjects between the ages of 18-55 who meet the criteria of one of the following four groups will be enrolled to measure serum and CSF Sema4A levels:

* Group 1: Newly diagnosed/untreated Relapsing MS patients (RMS)
* Group 2: Clinically stable RMS patients receiving disease modifying therapy (DMT)
* Group 3: RMS patients receiving DMT with breakthrough disease
* Group 4: Non-MS controls (patients without inflammatory CNS disease)

Participants will provide blood and CSF samples at baseline for Sema4A analysis. Follow up blood samples will be collected at 6 months and 12 months as part of lymphocyte subset analysis. Participation will end after 12 months of follow up.

The expected risks are related to blood draws and lumbar puncture. Lumbar puncture will be performed under fluoroscopy to decrease risks of pain from repeated needle punctures, injury from incorrect placement of the needle, and post puncture CSF leakage.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-55, inclusive at the time of consent
* Not pregnant at the time of the screening/baseline visit
* Able to understand the purpose, benefits, and risks of the study; willing and able to adhere to the study requirements; able and provide informed consent in English
* Meet the criteria of one of the four groups at the time of consent:

  * Group 1: subjects who have recently been diagnosed with MS, have had a clinical attack within the last 6 months, have not received steroids in the last 30 days, and have not started on a disease modifying therapy
  * Group 2: subjects with clinically stable relapsing MS, with no evidence of clinical relapse for at least the past 12 weeks, and have no gadolinium enhancing lesions on MRI in the prior 4 weeks, who are receiving a FDA-approved MS DMT
  * Group 3: subjects with relapsing MS on a FDA-approved DMT but with evidence of breakthrough disease, with a documented clinical relapse and/or gadolinium-enhancing lesion(s) on brain or spinal cord MRI taken within the 4 weeks
  * Group 4: subjects without evidence of inflammatory systemic or CNS disease, who require CSF removal for some other cause, such as for idiopathic intracranial hypertension or communicating hydrocephalus

Exclusion Criteria:

* There are no exclusion criteria for this study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Multiple sclerosis and non-MS controls
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-10-25 (Estimated); Study Completion 2023-10-25 (Estimated)

PRIMARY OUTCOMES:
Blood Serum Semaphorin 4A Levels | Baseline
  Measure blood serum semaphorin 4A levels at baseline
Cerebrospinal Fluid Semaphorin 4A Levels | Baseline
  Measure cerebrospinal fluid semaphorin 4A levels at baseline

SECONDARY OUTCOMES:
Correlation between Semaphorin 4A levels and Demyelination and Axonal Degeneration | 12 Months
  MRI will be performed at 6 months and 12 months to evaluate if there is a correlation between baseline semaphorin 4 A levels and demyelination and axonal degeneration.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Cohan, MD, PhD, Principal Investigator — Providence Health and Services
Locations (1):
- Providence St. Vincent Medical Center, Portland, Oregon, United States